CLINICAL TRIAL: NCT05320692
Title: A Phase III, Randomized, Open-Label, Multi-center Study of TACE Combined With Camrelizumab Plus Rivoceranib (Apatinib) or TACE Alone in Patients With Incurable Hepatocellular Carcinoma
Brief Title: A Study of TACE Combined With Camrelizumab Plus Rivoceranib (Apatinib) in Patients With Incurable Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-Ⅲ-336
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: This is a Randomized, Open-Label, Multi-center phase III clinical trial。
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): TACE Combined With Camrelizumab Plus Rivoceranib (Apatinib).
  Interventions: Drug: TACE+Camrelizumab+Apatinib mesylate
- Control group (Active Comparator): TACE Alone.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: TACE+Camrelizumab+Apatinib mesylate — TACE. Camrelizumab，200mg，iv，once every 3 weeks. Apatinib mesylate, 250 mg, administered orally once daily，once every 3 weeks.
  Arms: Treatment group
Procedure: TACE — TACE Alone.
  Arms: Control group

SUMMARY:
A study to evaluate efficacy and safety of transarterial chemoembolization (TACE) in combination with Camrelizumab and Rivoceranib (Apatinib) therapy in patients with incurable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study and sign informed consent.
2. Subjects diagnosed with HCC or clinically diagnosed with HCC by histopathology / cytology.
3. Baseline imaging examination has at least one measurable lesion.
4. Child-Pugh liver function rating was Grade A Within 7 days before randomization.
5. ECOG PS score within 7 days before randomization: 0 or 1. Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

1. Known hepatocholangiocarcinoma, sarcomatoid hepatocellular carcinoma, mixed cell carcinoma and lamellar cell carcinoma.
2. Subjects who are ready for or have previously received organ or allogeneic bone marrow transplantation.
3. Has any active autoimmune disease or a history of autoimmune disease and may relapse.
4. Suffering from hypertension and can not be well controlled by antihypertensive drugs.
5. With clinical symptoms or diseases of the heart that are not well controlled.
6. Previous or current central nervous system metastasis.
7. The subject has congenital or acquired immune deficiency (such as HIV infection).
8. Thrombotic or embolic events occurred within 6 months prior to the start of study treatment.
9. A history of gastrointestinal hemorrhage or a clear tendency to gastrointestinal bleeding within 6 months prior to the start of study treatment.
10. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months prior to the start of study treatment.
11. Severe, unhealed or cracked wounds and active ulcers or untreated fractures.
12. Known genetic or acquired bleeding or thrombotic tendencies.
13. Severe infection occurred within 4 weeks prior to the start of study treatment.
14. Received live attenuated vaccine treatment within 28 days prior to the start of study treatment.
15. Other investigational drugs were received within 28 days prior to the start of study treatment.
16. According to the assessment of investigator, the subject has other factors that may interfere with the results of the study or cause the forced termination of the study. Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by BIRC | approximately 5 years
  PFS is defined as the time from the date of randomization until the date of first objective disease progression or death (whichever occurs first).

SECONDARY OUTCOMES:
OS | approximately 5 years
  OS is defined as the time from the date of randomization until death due to any cause.
ORR | approximately 5 years
  ORR is defined as the percentage of participants in the analysis population who have a CR or PR.
DCR | approximately 5 years
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or SD.
DoR | approximately 5 years
  DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0 | approximately 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided